CLINICAL TRIAL: NCT03174418
Title: A Multicentre Prospective Study on the Role of Fluid Dynamics OCT-based REconstruction of Coronary Atherosclerosis in bifurcationS to Predict ouTcome
Brief Title: Fluid-dynamics in Bifurcation PCI
Acronym: FORECAST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesco Burzotta, MD, PhD, Catholic University of the Sacred Heart
Other Study IDs: 01012017
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Atherosclerosis, Coronary
Keywords: Optical coherence tomography; Percutaneous coronary interventions; Coronary atherosclerosis in bifurcations
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort A: Patients with bifurcated coronary lesions treated by percutaneous coronary interventions.
  Interventions: Procedure: Coronary angiography and optical coherence tomography
- Cohort B: Patients with untreated bifurcated coronary lesions.
  Interventions: Procedure: Coronary angiography and optical coherence tomography

INTERVENTIONS:
Procedure: Coronary angiography and optical coherence tomography — Coronary angiography and OCT images will be combined to obtain a three-dimensional model of the diseased coronary vessels that will be used to calculate the local blood flow patterns and the arterial time-averaged wall shear stress at the bifurcated lesion level

SUMMARY:
Investigator-initiated, international, multicentre, observational study with two cohorts.

The two study cohorts will be:

Cohort A: to understand if the local blood flow patterns (associated with low WSS), as evaluated by computational fluid dynamic tools from combined angiographic and OCT invasive images, may better predict the clinical outcome of patients with bifurcated coronary lesions treated by PCI.

Cohort B: to understand if the local blood flow patterns (associated with low WSS), as evaluated by computational fluid dynamic tools from combined angiographic and OCT invasive images, may better predict the clinical outcome of patients with sub-critical bifurcated lesions managed conservatively.

Coronary angiography and OCT images will be combined to obtain a three-dimensional model of the diseased coronary vessels that will be used to calculate the local blood flow patterns and the time-averaged WSS at the bifurcated lesion level by using computational fluid dynamics software.

Baseline (in patients both managed conservatively and treated by PCI) and post-PCI (in patients treated by PCI) images will be processed.

ELIGIBILITY:
Inclusion Criteria

* Patients with stable or unstable coronary artery disease;
* TIMI 3 on both MV and SB;
* MV visual diameter > 2.5 mm;
* SB visual diameter > 2.0 mm;
* Documentation of angiographically-critical (visually estimated percentage diameter stenosis ≥80% <100%) coronary lesion treated by PCI and underwent post-PCI OCT assessment or angiographically-intermediate (visually estimated percentage diameter stenosis ranging between 30-80%) lesion in the MV considered suitable for conservative management (myocardial revascularization not planned).

Exclusion Criteria

* Age < 18 years or impossibility to give informed consent.
* Female sex with child-bearing potential.
* Life expectancy of less than 12 months or factors making clinical follow-up difficult (no fixed address, etc.).
* Ascertained or suspected contraindications to prolonged (up to 6 month) double antiplatelet therapy.
* Known hypersensitivity to aspirin, heparin, contrast dye, sirolimus, everolimus, zotarolimus, cobalt, chromium, nickel, tungsten acrylic, and fluoro-polymers.
* Poor cardiac function as defined by left ventricular global ejection fraction ≤ 30%.
* Recent (< 48 hours) ST-segment elevation myocardial infarction.
* Severe myocardial hypertrophy (interventricular septum thickness > 15 mm, ECG Sokolow's criteria fulfilled).
* Severe valvular heart disease.
* Significant platelet count alteration (<100,000 cells/mm3 or > 700,000 cells/mm3).
* Gastrointestinal bleeding requiring surgery or blood transfusions within 4 previous weeks.
* History of clotting pathology.
* Advance renal failure with glomerular filtration rate < 30 ml/min (Cockcroft-Gault equation)
* Left main lesion.
* Target bifurcation located on a distal coronary segment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable or unstable coronary artery disease due to atherosclerosis involving a major bifurcation site, who undergo diagnostic or interventional invasive percutaneous coronary procedures with the use of optical coherence tomography (OCT) based on operator's choice.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Target bifurcation failure (TBF) | 1,6,12,18,24 and 36 months
  - Target bifurcated lesion-related major adverse coronary event (MACE) defined as the composite of:
  * cardiac death
  * myocardial infarction (MI) not clearly related with another vessel
  * target vessel revascularization (TVR)

SECONDARY OUTCOMES:
Target vessel failure | 1,6,12,18,24 and 36 months
  - In the absence of target bifurcated lesion-related MACE, target bifurcated lesion angiographic failure defined, in patients treated by PCI, as: > 50% restenosis on the main vessel (MV) or TIMI (Thrombolysis In Myocardial Infarction) flow < 3 on the side branch (SB) at angiography eventually performed during the clinical course.
Bifurcated lesion angiographic failure | 1,6,12,18,24 and 36 months
  * Cardiac death
  * MI
  * TVR
  * Definite or probable stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Burzotta, MD, Principal Investigator — Policlinico A. Gemelli. Università Cattolica del Sacro Cuore
Locations (1):
- Policlinico A. Gemelli. Università Cattolica del Sacro Cuore, Roma, Italy